CLINICAL TRIAL: NCT00239122
Title: Applicability of CBT to Unselected Mental Health Service Clients With Psychotic Disorders
Brief Title: Recovery Therapy Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: William Buckland Foundation (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E00013
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2005-10-14 (Estimated); Status verified 2005-10

CONDITIONS: Schizophrenia; Psychotic Disorders; Mood Disorders
Keywords: Cognitive Therapy; Psychotic Disorders; Treatment Outcome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mood Disorders | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Recovery Therapy (Cognitive Behaviour Therapy for psychosis)

SUMMARY:
This project will systematically apply a specialist version of Cognitive Behaviour Therapy (CBT), known as Recovery Therapy, to a random sample of patients with psychotic disorders. Previously, the therapy has been developed and efficacy established, but the extent of applicability to (unselected) mental health service patients is unknown. The main aim is to establish the extent to which this therapy is acceptable and effective for mental health service clients. A secondary aim is to develop guidelines for the conduct of such therapy in public mental health settings.

ELIGIBILITY:
Inclusion Criteria:

* acceptance by the participating Community Mental Health Services for case management
* a preliminary DSM-IV diagnosis of schizophrenia, schizoaffective disorder, mood disorder with psychotic features, or delusional disorder
* a recovery "need" in one of the areas addressed by the therapy

Exclusion Criteria:

* a preliminary DSM-IV diagnosis of brief psychotic disorder, drug-induced psychosis, mood disorder without hallucinations or delusions, or any other disorder (eg. personality disorder, PTSD) even where psychotic features are/have been present
* non-English speaking
* comorbid intellectual disability

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94
Dates: Start 2000-06; Study Completion 2004-02

PRIMARY OUTCOMES:
To determine the applicability of cognitive behaviour therapy for psychosis in the "real world" setting of ordinary mental health services

SECONDARY OUTCOMES:
To establish rates of uptake of Recovery Therapy amongst clients at a community mental health service
To establish effectiveness of therapy in clients who received a defined length of therapeutic contact (12-24 sessions)
To identify factors predicting uptake and effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: John Farhall, BA(Hons), MA, Principal Investigator — LaTrobe University, NorthWestern Mental Health
Locations (2):
- Australia (2):
  - Whittlesea Community Mental Health Service, Epping, Victoria
  - Darebin Community Mental Health Service, Preston, Victoria